CLINICAL TRIAL: NCT00287755
Title: Chemosensitivity Test to Evaluate the Effect of Adjuvant Cancer Chemotherapy (S-1) After Gastric Surgery
Brief Title: Clinical Trial of Chemosensitivity Test
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Japan Clinical Cancer Research Organization (Other)
Collaborators: Kitasato University (Other)
Responsible Party: Tetsurou Kubota / Professor, Center of Comprehensive and Advanced Medicine, Keio University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: JACCRO GC-04; GC-04
Record Dates: First submitted 2006-02-03; First posted 2006-02-07 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; S-1; chemosensitivity; adjuvant
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1 — S-1 capsule at a dose of 80 mg/m2 b.i.d. for 4 weeks followed by 2 weeks rest.

SUMMARY:
To evaluate the usefulness of chemosensitivity test in evaluating the appropriate adjuvant cancer chemotherapy after gastric surgery

DETAILED DESCRIPTION:
Patients: clinical Stage III gastric cancer patients. Informed consent will be obtained before surgery. Eligible patients: surgical Stage II, IIIA and IIIB gastric cancer patients. Chemosensitivity test: The surgical specimen will be sent Mitsubishi BCL, Co. Ltd. to be tested by CD-DST chemosensitivity test and RT-PCR for thymidylate synthetase and dihydropyrimidine dehydrogenase mRNA. The test results will be blinded for the doctors on duty.

Treatment: All the patients will be treated with S-1 at a dose of 80 mg/m2 b.i.d. for 4 weeks followed by 2 weeks rest. The treatment will be continued until the recurrence or 1 year after operation.

Primary endpoint: 3-years disease-free survival rate Secondary endpoint: 3-years overall survival rate and side effect (CTCAE v3.0) Evaluation of chemosensitivity test: The cutoff condition will be determined based on the accumulated data of CD-DST and mRNAs.

Hypothesis: The responder detected by CD-DST and/or TS, DPD mRNA will have a favorable survival outcome comparing with resistant cases.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven gastric cancer
* PS (ECOG) 0 or 2
* D2 dissection, curability B or more
* surgical Stage IIIA and IIIB
* negative peritoneal cytology
* no previous radiotherapy, chemotherapy and hormone therapy
* possible peroral intake at 6 POW
* no severe surgical complication
* normal bone marrow, liver and renal function
* complete chemosensitivity test
* written informed consent

Exclusion Criteria:

* multiple cancer
* contraindication for S-1
* history of drug allergy (grade 3)
* severe complication
* watery diarrhea
* pregnant
* scirrhous gastric cancer
* the other patients who was judged as inadequate for trial by doctor on duty

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-03; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | at three years

SECONDARY OUTCOMES:
Side effect | During administration of drug

CONTACTS AND LOCATIONS:
Overall Officials: Tetsuro Kubota, Processor, Principal Investigator — Keio University Hospital
Locations (36):
- Japan (36):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Department of frontier surgery,Draduate school of medicine,Chiba University, Chiba, Chiba
  - Kyusyu University Faculty of Medical Sciences, Fukuoka, Fukuoka
  - Kyusyu Central Hospital of the Mutual Aid Association of Public School Teachers, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Gunma University Hospital, Maehashi, Gunma
  - Hakodate Goryoukaku Hopsital, Hakodate, Hokkaido
  - Hyogo Prefectural Awaji Hospital, Sumoto, Hyōgo
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Kanazawa Medical University Hospital, Kanazawa, Ishikawa-ken
  - Iwate Medical University Hospital, Morioka, Iwate
  - Department of surgical oncology and digestive surgery kagoshima university graduate school, Kagoshima, Kagoshima-ken
  - Nippon Medical School Second Hospital, Kawasaki, Kanagawa
  - St. Marianna University, School of Medicine, Kawasaki, Kanagawa
  - Kitazato University East Hospital, Sagamihara, Kanagawa
  - Faculty of Medical and Pharmaceutical Sciences Kumamoto University, Kumamoto, Kumamoto
  - Niigata Prefectural Cancer Center, Niigata, Niigata
  - Hirakata City Hospital, Hirakata, Osaka
  - Osaka Kita Japan Post Hospital, Osaka, Osaka
  - Osaka City University Graduate School of Medicine, Osaka, Osaka
  - Saiseikai Suita Hospital, Suita, Osaka
  - Osaka Medical College Hospital, Takatsuki, Osaka
  - Yao Municipal Hospital, Yao, Osaka
  - Saga Medical School Faculty of Medicine,Saga University, Saga, Saga-ken
  - Jichi Medical School Hospital, Shimono, Tochigi
  - Dokkyo University School of Medecine, Shimotsuga, Tochigi
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - Surugadai Nihon University Hospital, Chiyoda-ku, Tokyo
  - Tobu Chiiki Hospital, Katsushika-ku, Tokyo
  - Cancer Institute Hospital, Koto-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Nippon Medical School Tama Nagayama Hospital, Tama, Tokyo
  - Tottori University Faculty of Medicine, Yonago, Tottori
  - Kouseiren Takaoka Hospital, Takaoka, Toyama
  - Wakayama Prefectural Medical University Hospital, Wakayama, Wakayama
  - Kanagawa Prefectural Cancer Center, Kanagawa, Yokohama

REFERENCES:
- [Derived] Tanigawa N, Yamaue H, Ohyama S, Sakuramoto S, Inada T, Kodera Y, Kitagawa Y, Omura K, Terashima M, Sakata Y, Nashimoto A, Yamaguchi T, Chin K, Nomura E, Lee SW, Takeuchi M, Fujii M, Nakajima T. Exploratory phase II trial in a multicenter setting to evaluate the clinical value of a chemosensitivity test in patients with gastric cancer (JACCRO-GC 04, Kubota memorial trial). Gastric Cancer. 2016 Apr;19(2):350-360. doi: 10.1007/s10120-015-0506-z. Epub 2015 Sep 18. PMID 26385385